CLINICAL TRIAL: NCT00255697
Title: Quality of Life Study Registry for Persons With Cancer and Family Caregivers
Brief Title: Quality of Life of Older Patients Who Are Undergoing Treatment for Cancer and of Their Family Caregivers
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE8Z05; P30CA043703 (NIH); CASE8Z05 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Psychosocial Effects of Cancer and Its Treatment; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: psychosocial effects of cancer and its treatment; unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: psychosocial assessment and care — Patients undergo a 45-minute interview in person or by phone to provide demographic data and to complete quality of life questionnaires, including Functional Assessment of Cancer Therapy (FACT), Spiritual tool, Quality and Satisfaction with Treatment (QUEST), and Profile of Mood State (POMS), at baseline and at 3 and 12 months. Caregivers undergo a 20- to 30-minute interview in person or by phone to provide demographic data and complete quality of life questionnaires, including the Caregiver Reaction Assessment (CRA), Quest, and POMS, at baseline and at 3 and 12 months. Caregivers complete the Quality of Death and Dying (QODD) questionnaire 2-3 months after the patient's death.
Procedure: quality-of-life assessment — Patients undergo a 45-minute interview in person or by phone to provide demographic data and to complete quality of life questionnaires, including Functional Assessment of Cancer Therapy (FACT), Spiritual tool, Quality and Satisfaction with Treatment (QUEST), and Profile of Mood State (POMS), at baseline and at 3 and 12 months. Caregivers undergo a 20- to 30-minute interview in person or by phone to provide demographic data and complete quality of life questionnaires, including the Caregiver Reaction Assessment (CRA), Quest, and POMS, at baseline and at 3 and 12 months. Caregivers complete the Quality of Death and Dying (QODD) questionnaire 2-3 months after the patient's death.

SUMMARY:
RATIONALE: Studying quality-of-life in patients having cancer treatment and in their caregivers may help identify the intermediate- and long-term effects of treatment on patients with cancer and on their caregivers.

PURPOSE: This clinical trial is studying quality of life of older patients who are undergoing treatment for cancer and of their family caregivers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Obtain quality of life and psychosocial data from older patients who are undergoing treatment for cancer and from their family caregivers.

OUTLINE: This is a pilot, cross-sectional study.

Patients undergo a 45-minute interview in person or by phone to provide demographic data and to complete quality of life questionnaires, including Functional Assessment of Cancer Therapy (FACT), Spiritual tool, Quality and Satisfaction with Treatment (QUEST), and Profile of Mood State (POMS), at baseline and at 3 and 12 months. Caregivers undergo a 20- to 30-minute interview in person or by phone to provide demographic data and complete quality of life questionnaires, including the Caregiver Reaction Assessment (CRA), Quest, and POMS, at baseline and at 3 and 12 months. Caregivers complete the Quality of Death and Dying (QODD) questionnaire 2-3 months after the patient's death.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patient:

  * Confirmed diagnosis of any type of cancer
  * Undergoing cancer treatment at Ireland Cancer Center
* Caregiver:

  * Identified family caregiver of a patient diagnosed with cancer
* Patient and caregiver may participate regardless of whether the other person agrees to participate or not

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-3 (patient)

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Able to speak and comprehend English
* Cognitively competent to be interviewed (patient)

PRIOR CONCURRENT THERAPY: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 863 (Actual)
Dates: Start 2005-07; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Functional status by Karnofsky and ECOG at baseline, 3 months, and 1 year | at baseline, 3 months, and 1 year
Co-morbidities by Charlson at baseline | at baseline
Cognitive status by Short Orientation Concentration Memory Test at baseline, 3 months, and 1 year | at baseline, 3 months, and 1 year
Quality of Life (QOL) by SF-12 at baseline | at baseline
QOL and Symptoms by Functional Assessment of Cancer Therapy-General (FACT-G) at baseline, 3 months, and 1 year | at baseline, 3 months, and 1 year
Spirituality by Functional Assessment of Chronic Illness Therapy (FACIT)-Sp at baseline, 3 months, and 1 year | at baseline, 3 months, and 1 year
Social Support by Shortened Social Support Scale at baseline, 3 months, and 1 year | at baseline, 3 months, and 1 year
Satisfaction with care by FACIT-TS-PS at 3 months and 1 year | at 3 months and 1 year
Mood state by Profile of Mood States at baseline, 3 months, and 1 year | at baseline, 3 months, and 1 year
Optimism by Life Orientation Test at baseline | at baseline
Caregiver Burden by Caregiver Reaction Assessment at baseline, 3 months, and 1 year | at baseline, 3 months, and 1 year

SECONDARY OUTCOMES:
Trends over time (mood state, satisfaction, symptoms, QOL, caregiver burden, and cognitive status) for patient and caregiver by the tools listed above at 3 months and 1 year | at 3 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Daly, PhD, RN, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States